CLINICAL TRIAL: NCT06845085
Title: Re-ablation of Persistent Atrial Fibrillation: a Randomized Study, Evaluating Vein of Marshall Ethanol Ablation in Combination With Block of Mitral and Tricuspid Isthmuses and Dome Line
Brief Title: Re-ablation of Persistent Atrial Fibrillation
Acronym: Re-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Karolinska University Hospital (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Peter Lukac, Consultant, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-10-72-153-24
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: Persistent atrial fibrillation; Radiofrequency ablation; Pulsed field ablation; Vein of Marshall alcohol ablation; Cavotricuspid isthmus line; Mitral isthmus line; Dome line; Pulmonary vein re-isolation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vein re-isolation plus VOM ablation and block of mitral and tricuspid isthmuses and dome line (Experimental): pulmonary vein re-isolation plus Vein of Marshall ethanol ablation in combination with block of mitral and tricuspid isthmuses and dome line
  Interventions: Procedure: Intervention
- vein re-isolation (Active Comparator): pulmonary vein re-isolation
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Intervention — pulmonary vein re-isolation plus Vein of Marshall ethanol ablation in combination with block of mitral and tricuspid isthmuses and dome line
  Arms: vein re-isolation plus VOM ablation and block of mitral and tricuspid isthmuses and dome line
Procedure: Control — pulmonary vein re-isolation
  Arms: vein re-isolation

SUMMARY:
Pulmonary vein re-isolation plus Vein of Marshall ethanol ablation in combination with block of mitral and tricuspid isthmuses and dome line will be compared to pulmonary vein re-isolation alone in patients undergoing re-ablation for persistent atrial fibrillation in this investigator initiated, randomized, patient-assessor blinded multicenter trial. Patients are followed with standard ECG at 3 months, with standard ECG, 5-days' ECG monitoring and quality of life assessment after 12 months, with standard ECG and quality of life assessment after 24 months, through patient files at 60 months after the ablation.

Primary endpoint: Change in AFEQT score between baseline and 12 months.

DETAILED DESCRIPTION:
This study is a prospective, patient and assessor blinded, 1:1 randomized superiority trial.

Consecutive patients referred for re-ablation of symptomatic PsAF after previous PVI will be included. All preoperative procedures will be conducted according to the department's standard operational procedures for AF ablation. In all patients, an electro anatomical map (CARTO™, Biosense Webster, Diamond Bar, CA, or EnSite X™, Abbott Laboratories, Abbott Park, IL) of the LA with a multipolar mapping catheter (PENTARAY™ or OCTARAY™, Biosense Webster, Diamond Bar, CA, or Advisor™ HD Grid, Abbott Laboratories, Abbott Park, IL) will be constructed and reconnection of PVs will be assessed in sinus rhythm. If reconnection is present, re-PVI will be performed and confirmed with the multipolar mapping catheter. Patients in atrial fibrillation will undergo cardioversion to sinus rhythm prior to mapping. After mapping and confirming isolation of the PVs, patients will be randomized using the Redcap Database software to intervention or control. The intervention group will undergo VOM ethanol ablation including supplementary LA and coronary sinus ablation, if needed to achieve mitral isthmus block plus creation of dome line and cavotricuspid isthmus (CTI) block. VOM ablation, mitral and CTI ablation and dome line will not be performed in control group and patients in control group will undergo no further ablation. The energy source used will be radiofrequency ablation or pulsed field ablation, at the discretion of the physician. However, radiofrequency should be preferred near coronary arteries. For dome line, focal PFA is preferred. All post-procedural work-up and follow-up will be the same for both randomization groups and assessment of outcomes will be performed by personnel blinded to randomization.

Patients are followed with standard ECG at 3 months, with standard ECG, 5-days' ECG monitoring and quality of life assessment after 12 months, with standard ECG and quality of life assessment after 24 months, through patient files at 60 months after the ablation.

Primary endpoint: Change in AFEQT score between baseline and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Previous pulmonary vein isolation for atrial fibrillation
* Indication for catheter ablation with at least two episodes of symptomatic PsAF during the last 12 months
* Age > 18 years
* Expected survival > 12 months
* Able to provide informed consent

Exclusion Criteria:

* Previous extrapulmonary atrial ablation other than cavotricuspid isthmus line, roof- or dome line or posterior wall isolation/ablation
* Atypical atrial flutter in addition to atrial fibrillation
* Atrial fibrillation secondary to a transient abnormality
* Uncontrolled hypertension
* Acute coronary syndrome, cardiac surgery, or TIA/stroke within the last 3 months
* Planned cardiac surgery within 1 year
* Dialysis or severe renal failure
* Active substance or alcohol abuse (>14 units/week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Change in Atrial fibrillation effect on quality of life (AFEQT) score | between baseline and 12 months
  A score with a scale from 0 to 100. The higher score signifies less disability

SECONDARY OUTCOMES:
Freedom from documented atrial arrhythmia | 12, 24 and 60 months
  As documented on a standard ECG or Holter, after 3 months blanking period, on or off antiarrhythmic drugs
Freedom from documented persistent atrial arrhythmia | at 12 and 24 months and 5 years
  duration 7 days or longer or cardioverted, after 3 months blanking period, on or off antiarrhythmic drugs
Freedom from direct-current cardioverted atrial arrhythmia | at 12 and 24 months and 5 years
  after 3 months blanking period, on or off antiarrhythmic drugs
Number of direct current-cardioversions and sustained atrial arrhythmia episodes | at 12 and 24 months and 5 years
  after 3 months blanking period, on or off antiarrhythmic drugs
Freedom from accepted chronic atrial fibrillation | at 12 and 24 months and 5 years.
  i.e. when cardioversion is not considered or indicated
Freedom from re-ablation procedure | at 12 and 24 months and 5 years.
  reablation procedure because of atrial arrhythmia
Change in Atrial fibrillation effect on quality of life (AFEQT) score | between baseline and 24 months and between baseline and 5 years.
  A score with a scale from 0 to 100. The higher score signifies less disability

CONTACTS AND LOCATIONS:
Locations (3):
- Department of Cardiology, Aarhus University Hospital, Århus N, Danmark, Denmark
- Department of Cardiology, Leiden University Medical Center, Leiden, Netherlands
- Department of Cardiology, Karolinska University Hospital, Stockholm, Stockholm, Sweden

DOCUMENTS (1):
  • Study Protocol (2025-01-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT06845085/Prot_000.pdf